CLINICAL TRIAL: NCT04951349
Title: Phase 2b Clinical Trial to Evaluate the Tolerability and Efficacy in Reducing the Nasal Viral Load of SARS-CoV-2 of Benzalkonium Chloride 0.0065% (GX-03), in the Form of Nasal Ointment, in Patients Infected With COVID -19, and Evaluation of Its Tolerability in Health Care Providers, as a Preventive of Nasal Colonization, Complementary to Personal Protective Equipment
Brief Title: Safety and Efficacy of Intranasal Application of GX-03 as a Treatment and Prevention for COVID-19.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Turn Therapeutics (Industry)
Collaborators: Gorgas Memorial Institute for Health Studies (Unknown); Hospital Santo Tomas (Other); Hospital Modular - Covid-19 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GX-03 for COVID-19
Record Dates: First submitted 2021-06-30; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Two part study with four total arms. Parts: Health care providers and CV-19 infected patients. Arms: Interventional and placebo in each of the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment of hospitalized patients with laboratory-confirmed COVID-19 (Experimental): Hospitalized patients with laboratory-confirmed COVID-19 using GX-03 administered intranasally TID for 5 days.
  Interventions: Drug: GX-03
- Placebo Treatment of hospitalized patients with laboratory-confirmed COVID-19 (Placebo Comparator): Hospitalized patients with laboratory-confirmed COVID-19 using placebo (petrolatum emulsion) administered intranasally TID for 5 days.
  Interventions: Drug: Petrolatum ointment
- Prevention of SARS-COV-2 in Health Care Providers (Experimental): Health care providers with laboratory-confirmed negative COVID-19 using GX-03 administered intranasally TID for 10 days.
  Interventions: Drug: GX-03
- Placebo Prevention of SARS-COV-2 in Health Care Providers (Placebo Comparator): Health care providers with laboratory-confirmed negative COVID-19 using placebo (petrolatum emulsion) administered intranasally TID for 10 days.
  Interventions: Drug: Petrolatum ointment

INTERVENTIONS:
Drug: GX-03 — Same dosage used in Bactroban Nasal studies.
  Other Names: Hexagen Antimicrobial
  Arms: Prevention of SARS-COV-2 in Health Care Providers; Treatment of hospitalized patients with laboratory-confirmed COVID-19
Drug: Petrolatum ointment — Viscous ointment similar in form to study drug.
  Other Names: Placebo
  Arms: Placebo Prevention of SARS-COV-2 in Health Care Providers; Placebo Treatment of hospitalized patients with laboratory-confirmed COVID-19

SUMMARY:
Phase 2b clinical trial to evaluate the safety and efficacy of intranasal application of GX-03 as a treatment and prevention for COVID-19.

DETAILED DESCRIPTION:
Phase 2b clinical trial to evaluate the safety and efficacy of intranasal application of GX-03 as a treatment and prevention for COVID-19. Patients hospitalized with a diagnosis of mild to moderate COVID-19 will be evaluated for a period of five days. Participating health care providers will be evaluated for a period of ten days. Swab samples will be collected from the right and left anterior nostrils at the beginning of the study, as well as three times per day in the treatment arm for five days. Swab samples will be collected from the right and left anterior nostrils at the beginning and end of the prevention arm. Samples will be subjected to biomolecular tests and viral cultures to assess positivity and disease progression. Safety will be evaluated through standard measures of erythema and edema in the nasal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18-65 hospitalized with SARS-CoV-2, diagnosed by a positive nasal or nasopharyngeal swab

  2. Men or women who are not pregnant, not breastfeeding, postmenopausal, naturally or surgically sterile, or who agree to use effective contraception during the course of the study. A postmenopausal patient is defined as at least 12 12 months of natural spontaneous amenorrhea or at least 6 weeks after surgical menopause (bilateral oophorectomy).

  3. Women of childbearing age who use one of the following acceptable contraceptive methods can be included in the study:

Surgical sterilization (hysterectomy and/or bilateral oophorectomy);

Surgical sterilization (surgical bilateral tubal ligation at least 6 weeks prior to screening); Intrauterine device (IUD) placed at least 3 months prior to detection; Abstinence (not having heterosexual sex);

Barrier method (condom or diaphragm) with spermicide for at least 14 days before selection and until completion of the study;

Stable hormonal contraceptive for at least 3 months prior to selection and until completion of the study

4. Patients capable of understanding and providing signed informed consent.

Exclusion Criteria:

1. SARS-CoV-2 positive patients on a ventilator.
2. Patients with any open wounds, injuries, inflammation, erythema, or infection (other than COVID-19) affecting the nasal passages, nose, upper lip, and the area of skin around the nose, including herpes simplex lesions.
3. Patients with a history of abnormal bleeding, bruising, frequent nosebleeds, or those diagnosed with von Willebrand disease.
4. Patients with nasal polyps or significant anatomical nasal abnormalities.
5. Patients with a history of nasal surgery, including cauterization, in the last 6 months.
6. Patients who currently have or have ever had a nose or septum piercing
7. Patients treated with antiviral medications in the past 7 days
8. Known allergy or history of significant adverse reactions to benzalkonium chloride or related compounds, or to any of the excipients.
9. Known or suspected pregnancy, pregnancy planned during the study period, or breastfeeding.
10. Clinically significant mental illness (to be determined by the investigator)
11. Recent history of (last 12 months) or strong potential for alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz of beer, 5.0 oz of wine, or 1.5 oz of distilled spirits)
12. Exposure to any agents being researched within 30 days prior to admission to the study.
13. Prior enrollment in this study
14. If the patient has a condition that the investigator believes would interfere with their ability to give informed consent or comply with study instructions, or that could confuse the interpretation of study results or put the patient at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Reduction of 60% in viral load from baseline | 5 days
  Time to achieve a 60% reduction in viral load from baseline.
Primary Safety analysis | 5-10 days
  To evaluate the incidence rate(s) of non-serious and serious adverse events associated with administration of the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Sandoval, MD, Principal Investigator — Medical Corps of Punta Pacifica Hospital
Locations (3):
- Panama (3):
  - Gorgas Memorial Research Hospital, Panama City
  - Hospital Modular COVID-19, Panama City
  - Hospital Santo Tomas, Panama City

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: Within 30 days of announcement of study completion.
Access Criteria: By official request for qualified use.